CLINICAL TRIAL: NCT06788418
Title: Comparative Study of SMILE, ICL, and Wavelight Plus Alcon Technologies in Myopia Correction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Visionly Plus Eye Hospital (Other)
Collaborators: High Myopia Control Alliance (HIMALAYA) (Unknown); Beijing New Vision Eye Hospital (Unknown); Shanghai Parkway Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Himalaya202501
Record Dates: First submitted 2025-01-22; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Myopia
Keywords: myopia; Small Incision Lenticule Extraction; Implantable Collamer Lens; Wavelight Plus Alcon system; vision
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SMILE Group (Experimental): Standard Small Incision Lenticule Extraction (SMILE) procedure using VisuMax laser
  Interventions: Procedure: SMILE
- ICL group (Experimental): Implantable Collamer Lens (ICL) implantation using the STAAR Surgical Visian ICL
  Interventions: Procedure: ICL
- Wavelight Plus Alcon Group (Experimental): Laser vision correction using the Wavelight Plus Alcon system
  Interventions: Procedure: Wavelight Plus Alcon system

INTERVENTIONS:
Procedure: Wavelight Plus Alcon system — Wavelight Plus Alcon system guided surgery for myopia
  Other Names: Small Incision Lenticule Extraction; Implantable Collamer Lens
  Arms: Wavelight Plus Alcon Group
Procedure: SMILE — Small Incision Lenticule Extraction surgery for myopia
  Arms: SMILE Group
Procedure: ICL — Implantable Collamer Lens surgery for myopia
  Arms: ICL group

SUMMARY:
Myopia is a prevalent refractive error with significant lifestyle impact. While traditional SMILE (Small Incision Lenticule Extraction) and ICL (Implantable Collamer Lens) surgeries are standard options, the advent of the Wavelight Plus Alcon system presents a promising new technique. This trial aims to evaluate the safety, efficacy, and patient satisfaction across these methods.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-40 years
* Spherical equivalent of -1.00 to -10.00 D
* Stable refraction for at least 12 months
* Informed consent provided

Exclusion Criteria:

* Other ocular pathologies
* Previous refractive surgery
* Pregnancy or nursing
* Autoimmune or connective tissue disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Vision at 12 months post-surgery | From the day of surgery through to the 12-month post-operative follow-up
  Uncorrected distance vision (UDVA) at 12 months post-surgery

SECONDARY OUTCOMES:
Change in spherical equivalent at 12 months post-surgery | From the day of surgery through to the 12-month post-operative follow-up
  Change of the spherical equivalent at 12 months post-surgery

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing New Vision Eye Hospital, Beijing
  - Beijing Visionly Plus Eye Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2025-January 2027

REFERENCES:
- [Background] Meng ZY, Yang L, Zhou P. Femtosecond laser versus manual clear corneal incision in implantable collamer lens surgery. Sci Rep. 2025 Jan 7;15(1):1086. doi: 10.1038/s41598-024-81477-w. PMID 39774960